CLINICAL TRIAL: NCT05319457
Title: Testing Radon Com Methods: Clinical Trial Smartphone App vs Print Brochures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Dakota (Other)
Responsible Party: Principal Investigator, Soojung Kim, Associate Professor, University of North Dakota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTR radon PCF
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Print brochures (Placebo Comparator): Participants assigned to the print brochure group will receive three educational print brochures about radon published by EPA via postal mails for three months (one per each month).
  Interventions: Other: Print brochure
- The radon app (Experimental): Participants assigned to the radon app group will be asked to use the radon app for three months where they will be exposed to mobile friendly educational content that is repurposed from educational print brochures about radon published by EPA.
  Interventions: Other: The radon app

INTERVENTIONS:
Other: The radon app — Participants will be asked to use the radon app.
  Arms: The radon app
Other: Print brochure — Participants will receive print brochures.
  Arms: Print brochures

SUMMARY:
The purpose of this research study is to compare the effectiveness of radon information delivered via the radon app vs. a traditional approach (printed brochure). The prevalence of exceptionally high levels of residential radon in ND, coupled with public's poor understanding of this hazard, is a critical public health problem.

ELIGIBILITY:
Inclusion Criteria:

* The principal eligibility criterion is that participants own a smartphone.

Exclusion Criteria:

* The principal exclusion criterion is previous testing for radon within the past two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Ordering a free radon test kit | Through the study completion - 3 months
  The rate at which participants order a free radon test kit
Using the radon test kit | Through the study completion - 3 months
  The rate at which participants use the radon test kit to test their houses
Change from baseline radon knowledge at 3 months | Change from baseline knowledge level to the completion of study at 3 months
  Participants' knowledge about radon and its dangers, how to protect themselves from radon, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Soojung Kim, Study Director — University of North Dakota; Gary G Schwartz, Principal Investigator — University of North Dakota
Locations (1):
- University of North Dakota, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim S, Scheffer-Wentz H, Klug MG, Schwartz GG. Comparing Communication Methods to Increase Radon Knowledge and Home Testing: A Randomized Controlled Trial in a High-Radon City. Int J Environ Res Public Health. 2023 Apr 25;20(9):5634. doi: 10.3390/ijerph20095634. PMID 37174154